CLINICAL TRIAL: NCT03725306
Title: Librata Endometrial Ablation Device Treatment to Reduce Menstrual Blood Loss
Acronym: LEADER
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: LiNA Medical (Industry)
Collaborators: Syntactx (Network); West Virginia University, Pathology Laboratory for Translational Medicine (Unknown); Infinite Clinical Research, S.A. de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LEADER NA
Record Dates: First submitted 2018-10-29; First posted 2018-10-31 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Menorrhagia; Heavy Menstrual Bleeding
Keywords: Heavy Menstrual Bleeding; Endometrial Ablation
MeSH Terms: conditions — Menorrhagia

STUDY DESIGN:
Intervention Model Description: Objective Performance Criterion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Librata (Experimental): Librata Endometrial Ablation Device
  Interventions: Device: Librata

INTERVENTIONS:
Device: Librata — Hyperthermic endomyometrial treatment via Librata catheter and balloon device

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of the endometrial ablation device Librata in reducing menstrual blood loss at 12 months post-treatment when used in pre-menopausal women with menorrhagia due to benign causes for whom childbearing is complete.

DETAILED DESCRIPTION:
Menorrhagia is ovulatory (cyclic), heavy bleeding, that should be treated when it interferes with quality of life or causes anemia. It is a common problem and it is estimated that 5% of women aged 30 to 49 seek referral for evaluation and treatment. No structural cause is found in the majority of women with menorrhagia and treatment intends to reduce blood loss and improve quality of life.

First line treatment is medical therapy with hormonal therapy using either the combined contraceptive pill or the levonorgestrel-releasing intrauterine system. These treatments are not suitable for all women and indeed some women may not find them acceptable. For these women, surgical management is then offered with either endometrial ablation or hysterectomy.

The primary objective of this study is to evaluate the clinical success defined as a reduction of menstrual bleeding, defined as a score of 75 or less or 50% reduction from baseline on the Menstrual Pictogram scoring diary at 12 months post-treatment. Additionally, a secondary objective is to determine the primary safety incidence of serious adverse events (SAEs) by 12 months.

The study is designed as a prospective, multi-center, single-arm, controlled trial to demonstrate that the percentage of subjects with reduction in menstrual bleeding at 12 months is significantly greater than 66%. A total of 200 subjects will be enrolled.

The study population will include pre-menopausal women, aged 25-50 with a history of menorrhagia due to benign causes for whom childbearing is complete.

ELIGIBILITY:
Candidates for this study must meet ALL of the following criteria:

* Refractory menorrhagia with no organic cause
* Female subject from (and including) age 25 to 50 years
* Uterine sound measurement ≥6.0 cm to ≤ 10.0cm (external os to fundus).
* A minimum menstrual blood loss

  * for subjects not using medical therapy, a Menstrual Pictogram(MP) score of ≥150 for two baseline cycles within three months prior to treatment OR
  * MP score ≥150 for one month for women who either had

    * at least 3 prior months documented failed medical therapy; or
    * had a contraindication to medical therapy; or
    * refused medical therapy
* Premenopausal at enrollment as determined by FSH measurement ≤ 40 IU/L
* Not pregnant and no desire to conceive at any time
* Subject agrees to use a reliable form of contraception. If a hormonal birth control method is used, the subject must have been on said method for ≥ 3 months prior to enrollment and agrees to remain on the same hormonal regimen through their study participation.
* Able to provide written informed consent using a form that has been approved by the reviewing IRB/EC
* Subject agrees to follow-up visits and data collection requirements
* Subject who is literate or demonstrates an understanding on how to use the Menstrual Pictogram (MP) diary 4.1.1. EXCLUSION CRITERIA

To be enrolled, candidates should NOT meet any exclusion criterion:

* Pregnancy or subject with a desire to become pregnant
* Endometrial hyperplasia as confirmed by histology
* Presence of active endometritis
* Active pelvic inflammatory disease
* Active sexually transmitted disease (STD), at the time of ablation.

  o Note: Treatment of STD documented in the chart serves as sufficient evidence of infection resolution. Subject may be considered for study enrollment.
* Presence of bacteremia, sepsis, or other active systemic infection
* Active infection of the genitals, vagina, cervix, uterus or urinary tract at the time of the procedure
* Known/suspected gynecological malignancy within the past 5 years
* Known clotting defects or bleeding disorders
* Untreated/unevaluated cervical dysplasia (except CIN I)
* Known/suspected abdominal/pelvic cancer
* Prior uterine surgery (except low segment cesarean section) that interrupts the integrity of the uterine wall (e.g., myomectomy or classical cesarean section)
* Previous endometrial ablation procedure
* Currently on medications that could thin the myometrial muscle, such as long-term steroid use (except inhaler or nasal therapy for asthma)
* Currently on anticoagulants
* Abnormal or obstructed cavity as confirmed by transvaginal ultrasound +/- hysteroscopy - specifically:

  1. Septate or bicornuate uterus or other congenital malformation of the uterine cavity
  2. Submucosal fibroids (grade 0-2) which protrude >1cm into the uterine cavity
  3. Polyps >2 cm in maximum diameter
  4. Any intramural myoma > 3 cm or which distorts the uterine cavity
* Presence of an intrauterine device (IUD) which the subject unwilling to have removed at the time of the operative visit
* Presence of an implanted contraceptive device (e.g. Essure or Adiana).
* Subject not currently on hormonal birth control therapy and unwilling to use a non-hormonal birth control post-ablation
* Subject wanting concomitant hysteroscopic sterilization
* Subject who is within 6-weeks post-partum
* Any general health condition which, in the opinion of the Investigator, could represent an increased risk for the subject
* Any subject who is currently participating in the primary endpoint phase of an on-going investigational drug or device study or intends future participation in any other research of an investigational drug or device during the primary endpoint phase of this study

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pre-menopausal women for whom childbearing is complete
Enrollment: 200 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Menstrual Bleeding | 12 months post-treatment
  Clinical success defined as a reduction of menstrual bleeding, defined as a score of 75 or less or 50% reduction from baseline on the Menstrual Pictogram scoring diary.
Incidence of serious adverse events (SAEs). | 12 months post-treatment
  The primary safety endpoint

SECONDARY OUTCOMES:
Changes in Quality of Life | 12 months
  Responses from quality of life questionnaires
Procedure Time | During procedure
  Librata ablation procedure time
Menstrual Blood Loss | 3, 6, 12, 24 and 36 months
  Menstrual blood loss assessment
Rates of Re-Intervention | Month 12
  Rate of repeat ablation and/or hysterectomy surgery
Incidence of Unanticipated Adverse Device Effects (UADEs) | Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Claude Fortin, MD, Principal Investigator — LaSalle, QC

IPD SHARING:
Plan to Share IPD: No